CLINICAL TRIAL: NCT05996653
Title: A Multi-institutional Observational Study of CEST Imaging in Low-grade Glioma
Brief Title: CEST in Low-grade Glioma Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. MaryJane Lim Fat, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5396
Record Dates: First submitted 2023-07-06; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Low-grade Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ST-MRI scans (Other): All patients will undergo Saturation Transfer (ST)-MRI during their standard of care imaging visits (or within 14 days of their standard MRI).
  Interventions: Diagnostic Test: Saturation Transfer (ST)-MRI

INTERVENTIONS:
Diagnostic Test: Saturation Transfer (ST)-MRI — Non-contrast magnetic resonance imaging "Saturation Transfer" scans consisting of magnetization transfer (MT) and chemical exchange saturation transfer (CEST)

SUMMARY:
Low grade gliomas (LGGs) are malignant, infiltrative and incurable brain tumours that typically present in the younger population. This project proposes to use non-contrast metabolic "Saturation Transfer" (ST)-MRI to evaluate LGG tumour progression and aims to predict early changes in LGG. Early identification of LGG patients whose tumours will progress will permit early interventions. ST-MRI does not involve any intravenous injection of contrast and which acquires metabolic information not seen by standard MRI.

DETAILED DESCRIPTION:
Please see trial details below:

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 12 years of age;
2. Diagnosed with:

   1. Cohort A (pre-surgical): Suspected LGG (oligodendroglioma or astrocytoma), based on any combination of histological, molecular, radiological, and/or clinical findings; or
   2. Cohort B (post-surgical): IDH1/2-mutant or IDH-wildtype (WT) low-grade glioma candidate for observation
3. No contraindications to MRI;
4. eGFR > 30 ml/min;
5. No prior chemotherapy or radiation therapy;
6. No need for upfront treatment (surgery, chemotherapy, and/or radiation therapy)
7. Followed at either Sunnybrook Health Sciences Centre or at St Michael's Hospital

Exclusion Criteria:

1. Need for upfront post-surgical treatment with either chemotherapy and/or radiation therapy
2. Pregnancy

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-12 (Actual); Primary Completion 2028-08-12 (Estimated); Study Completion 2028-08-12 (Estimated)

PRIMARY OUTCOMES:
The time-to-progression as measured by Saturation Transfer (ST)-MRI (based on a change in volume or parameter value of over 10%) relative to the time-to-progression as measured by standard MRI using RANO-LGG. | Up to 6 years, from date of initial (ST)-MRI scan until the date of progression
  Time-to-progression refers to clinical progression of a low-grade glioma to a higher tumour grade.

SECONDARY OUTCOMES:
Accuracy of Saturation Transfer (ST)-MRI for detecting progression (based on a change in volume or parameter value of over 10%). | Up to 6 years, from date of initial (ST)-MRI scan until the date of progression
  The accuracy will be measured based on Saturation Transfer (ST)-MRI alone without standard MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Greg J Stanisz, PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario